CLINICAL TRIAL: NCT06295081
Title: TREAT Study - Improving the Interpretation of Troponin Concentrations Following Exercise and Their Clinical Significance
Acronym: TREAT
Status: Active, not recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL79864.091.22; 112927 (Other: RadboudUMC)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; exercise; athlete; troponin; radiology; biomarker
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for assessment of biomarker concentrations in serum and/or plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Walkers: Amateur athletes who perform a walking exercise with a minimum distance of 20 km
  Interventions: Other: Exercise exposure
- Runners: Amateur athletes who perform a running exercise with a minimum distance of 15 km
  Interventions: Other: Exercise exposure
- Cyclists: Amateur athletes who perform a cycling exercise with a minimum distance of 100 km
  Interventions: Other: Exercise exposure

INTERVENTIONS:
Other: Exercise exposure — Exercise is NOT part of our study protocol. Participants will voluntarily participate in a mass-participation exercise event (i.e. walking, cycling or running). Participation in this exercise event is voluntary and independent from participation in this study (i.e. participants would also take part in the exercise event if they did not participate in our study). Therefore, we do not consider the performed exercise an intervention or part of our study protocol. Hence, we consider our study design to be observational.
  Participants will perform exercise during a mass-participation exercise event, stratified for type of exercise (walking versus running versus cycling; n=500 each).
  The mass-participation exercise events have a sport-specific minimum distance of:
  a mass-participation exercise event with a:
  * Walking distance ≥20 km
  * Cycling distance ≥100 km
  * Running distance ≥15 km

SUMMARY:
The goal of this observational study is to learn about cardiac biomarker release following exercise in amateur athletes.

The main questions it aims to answer are:

Question 1: What are the reference values for exercise-induced cardiac troponin elevations following walking, cycling and running exercise? Hypothesis 1: We hypothesize that the exercise-induced cTn release is different following walking, cycling and running exercise. Therefore, we will establish reference values for post-exercise cTn concentrations across each of these sport types.

Question 2: Is the prevalence of (subclinical) coronary artery disease higher in individuals with high post-exercise cardiac troponin concentrations in comparison to individuals with low post-exercise cardiac troponin concentrations? Hypothesis 2: We hypothesize that athletes with the highest post-exercise cTn concentrations have a higher prevalence of coronary atherosclerosis compared to athletes matched for sex and age with the lowest post-exercise cTn concentrations.

Question 3: What is the association between post-exercise cardiac troponin concentrations and major adverse cardiovascular events (MACE) and mortality during long-term follow-up? Hypothesis 3: We hypothesize that post-exercise cTn concentrations beyond the 99th percentile are associated with an increased risk for MACE and mortality during follow-up.

This study consists of three phases:

Phase 1: two or three visits to the study location for (amongst other measurements) blood draws to assess cardiac troponin concentrations

Phase 2: CT scan of the heart in 10% of participants to assess the prevalence of (subclinicial) coronary artery disease.

Phase 3: longitudinal follow-up to assess the incidence of major adverse cardiovascular events and mortality during 20-year follow-up.

Participants will visit our study centre two, three or four times:

Visit 1: baseline measurements including height, weight, body composition and blood pressure will be obtained and a blood sample will be drawn.

Visit 2: a blood sample will be drawn and activity data will be obtained from participants' own sports watch or bike computer.

Optional visit 3: a blood sample will be drawn. Visit 4: 10% of participants will undergo a cardiac CT scan to assess the prevalence of (subclinical) coronary artery disease.

DETAILED DESCRIPTION:
For a detailed description, please see the attached study protocol under 'Documents'.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Participant of an affiliated mass-participation exercise event with a:

  * Walking distance ≥20 km
  * Cycling distance ≥100 km
  * Running distance ≥15 km
* Age: ≥ 40 and <70 years old
* Able to understand and perform study related procedures

For Phase 2 of the study (i.e. assessment of (sub)clinical coronary artery disease), the following additional criteria are present:

• Free from (known) cardiovascular diseases

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in Phase 2 of the study:

* Renal transplantation in the past
* Contrast nephropathy in the past
* estimated glomerular filtration rate (eGFR) < 30 ml/min
* Atrial fibrillation (heart rhythm disorder)
* Previous allergic reaction to iodine contrast
* Participation in other studies involving radiation
* Not willing to be informed about potential incidental findings from the CT-scan

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1500 Athletes will be recruited at mass-participation long-distance exercise events and stratified for type of sport (e.g. walking, cycling, running). Recruitment will take place via official websites/newsletters of the associated exercise events and social media channels.
  Our research has extensive experience performing studies in mass-participation exercise events, such as the Four Days Marches, Seven Hills Run, Eindhoven Marathon, Amsterdam Marathon, Maastricht Marathon in which we successfully included hundreds of participants. Therefore, we expect no difficulty to reach our target number of included participants.
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2044-07-01 (Estimated)

PRIMARY OUTCOMES:
High-sensitivity cardiac troponin I (hs-cTnI) | Within 5 days before exercise event, within 6 hours post-exercise cessation, 24-48 hours post-exercise cessation
  Concentrations of high-sensitivity cardiac troponin I (hs-cTnI) in plasma in ng/L
High-sensitivity cardiac troponin T (hs-cTnT) | Within 5 days before exercise event, within 6 hours post-exercise cessation, 24-48 hours post-exercise cessation
  Concentrations of high-sensitivity cardiac troponin T (hs-cTnT) in plasma in ng/L

SECONDARY OUTCOMES:
General CT scan data | within 3 months after inclusion
  CT scan date (dd-mm-yyyy); average heart rate during scan (bpm); total radiation dose (mSv); beta-blockers administration (yes/no, if yes: dose (mg)); nitro-glycerine administration (yes/no, if yes: dose (mg)); image quality (good/moderate/poor); FFR series obtained (yes/no, if yes: quality(good/moderate/poor)); incidental findings.
Coronary artery calcification score | within 3 months after inclusion
  Coronary artery calcium score [=CACS], per coronary artery or other (LM/LAD/LCX/RCA/RI/Aorta/Valves/Other) and total: lesion count (n); Agatston score (AU); volume (mm3); density (HU). Total CACS (AU); total volume (mm3); total density (HU); MESA percentile (%).
  LM: left main; LAD: left anterior descending; LCX: left circumflex; RCA: right coronary artery; RI: ramus intermedius; AU: Agatston units; HU: Hounsfield units; MESA: Multi-Ethnic Study of Atherosclerosis.
Coronary stenosis and plaque characteristics | within 3 months after inclusion
  Coronary stenoses, per segment (1-18): maximum stenosis degree (0%/1-24%/25-49%/50-69%/70-99%/100%/non-diagnostic/vessel absent); number of calcified plaques (n); number of partially calcified plaques (n); number of non-calcified plaques (n).
  Presence of myocardial bridging (yes/no); heart 'dominance' (PDA supplied by RCA/PDA supplied by LCX); room for general comments on CT scan.
  In general, not per segment: stenosis involvement score (n); stenosis severity score (n); plaque burden (P0/P1/P2/P3/P4); high-risk plaque features, per type [low attenuation plaque/positive remodelling/spotty calcification/napkin ring sign] (yes/no); modifiers, per modifier [non-diagnostic/having ≥high-risk plaque features/ischemia/exceptions including coronary artery dissection, anomalous origin of the coronary arteries, coronary artery (pseudo) aneurysm, vasculitis, coronary artery fistula, extrinsic coronary artery compression, arterio-venous malformation, other causes] (yes/no); CAD-RADS 2.0 score.
Computed tomography derived Fractional Flow Reserve | within 3 months after inclusion
  CT-derived FFR per coronary artery (LM/LAD/LCX/RCA): FFR at the beginning of vessel (ratio); FFR at 1.5 mm diameter of vessel or most distal evaluable part (ratio); FFR at 20 mm distal from stenosis (ratio).
  FFR signs for ischemia present [=FFR≤0.75] (yes/no); borderline ischemia [=FFR 0.76-0.80] (yes/no), non-ischemia [=FFR >0.80] (yes/no).
  FFR: fractional flow reserve
Incidence of mortality | 5 years after inclusion, 10 years after inclusion, 15 years after inclusion, 20 years after inclusion. Time-to-event: From the date of inclusion until the date of first documented date of death (from any cause), assessed up to 20 years after inclusion
  Incidence of mortality (yes/no), if yes: date of death (dd-mm-yyyy) and cause of death; cardiovascular death (yes/no).
Incidence of major adverse cardiovascular events | At 1/2/3/4/5/6/7/8/9/10/11/12/13/14/15/16/17/18/19/20 years after inclusion.Time-to-event: From the date of inclusion until the date of first documented major adverse cardiovascular event, assessed up to 20 years after inclusion.
  Incidence of MACE (yes/no), if yes: date, type of event (myocardial infarction/stroke/heart failure/revascularisation (both acute and elective)/sudden cardiac arrest), hospitalization (yes/no).
  MACE: major adverse cardiovascular events.

OTHER OUTCOMES:
Participant characteristics (personal info) | At day of inclusion
  Sex (male/female); name; e-mail address; phone number; place of residence; date of birth (dd-mm-yyyy); mass-participation sports event; distance (km).
  If included in the study: Participant identification number (TREAT…).
Participant characteristics (baseline measurements) | At day of inclusion
  Blood pressure: Systolic and diastolic blood pressure (mmHg) at rest; heart rate at rest (bpm).
  Anthropometry: Height (cm); weight (kg); BMI (kg/m2); body fat percentage (%); fat-free mass (kg ).
  BMI: body mass index;
Participant characteristics (Exercise characteristics): | Visit 2 (within 6 hours post-exercise cessation)
  Exercise type (walking/cycling/running); exercise distance (km); start and finish time (hh:mm); pause time (hh:mm); exercise duration (hh:mm); average speed (km/h); average speed (min/km); average heart rate (bpm).
  If used a sports watch or bike computer: .FIT-file or .CSV-file of activity.
Medical History questionnaire, part 1 (general info and cardiovascular complaints) | Within 1 week following inclusion
  General: level of education (primary education/preparatory vocational education/secondary vocational education/university of applied sciences/university bachelor/university master/PhD/other); ethnicity (Caucasian(European)/Afro-American/Asian/mixed/other); smoking (yes/no but I used to smoke/never); alcohol consumption (units/week); frequency of being active for ≥30 minutes (days/week); ever used performance-enhancing substances (yes/no, if yes: which substances).
  Cardiovascular complaints and/or procedures: cardiovascular complaints [e.g. dyspnoea, chest pain, fainting, palpitations] (yes/no); ever had coronary stenting or coronary artery bypass grafting (yes/no, if yes: reason of procedure, year and hospital where procedure was performed).
Medical History questionnaire, part 2 (diseases and/or conditions) | Within 1 week following inclusion
  Diseases and/or conditions (all yes/no, if yes, date of diagnosis (dd-mm-yyyy)): atherosclerosis; stroke/TIA/CVA; atrial fibrillation; COPD/lung diseases; embolism [anywhere other than lungs]; erectile disorders; intermittent claudication; myocardial fibrosis; fainting; conduction disorders; heart attack/myocardial infarction; heart failure; heart rhythm disorder; heart murmur; hypertrophic cardiomyopathy; lung embolism; kidney failure or kidney disorders; myocarditis; angina/chest pain; rheumatic disorders; diabetes mellitus; thrombosis; vascular dementia; hypertension; hypercholesterolaemia; hypotension; narrowed/occluded artery; dilation of artery [aneurysm], disease of lymph nodes or vessels, other diseases (yes/no, if yes: which disease and date of diagnosis (mm-yyyy).
Medical History questionnaire, part 3 (family history, COVID-19 info and medication use) | Within 1 week following inclusion
  Family history of cardiovascular diseases in 1st-degree family members before age 60 years: sudden death <50 years (yes/no); myocardial infarction or cardiac arrest (yes/no); coronary stenting or coronary artery bypass grafting (yes/no); stroke [cerebral infarction or haemorrhage] (yes/no); high cholesterol (yes/no); dilation of an artery [aneurysm] (yes/no); narrowing of an artery [stenosis] (yes/no, if yes: which artery (carotid/coronary/legs/other).
  COVID-19: had coronavirus infection (yes/no/probably, if yes or probably: date of infection (dd-mm-yyyy) and how the infection was diagnosed (PCR test/CT scan/antigen test/self-test/general practitioner or medical specialist diagnosed/I only have a suspicion that I had a coronavirus infection).
  Medication use: participant uses medication regularly in the last year (yes/no, if yes: name of drug, dose (mg), frequency (doses/day), comments) Other: room for further comments regarding health in general
Exercise History questionnaire, part 1 (exercise history, participation in endurance races and current training status) | Within 1 week following inclusion
  Lifetime exercise history (if multiple sports: the following data will be collected per sport discipline): sport discipline; age started (years); age quit (years); frequency (days/week); frequency (months/year); average duration of a session (minutes).
  Participation in endurance races (how often participated in the following races/events): Zevenheuvelenloop (n); half marathon (n); marathon (n); ultra marathon (n); Nijmegen Four Days Marches (n); Kennedy march [80 km] (n); cycling events ≥120 km (n); Alpe d'HuZes (n); triathlon sprint (n); triathlon quart or half (n); triathlon whole/Ironman (n); other endurance races.
  Current endurance activities (if multiple sports: the following data will be collected per sport discipline): sport discipline; age started (years); age quit (years); frequency (days/week); frequency (months/year); average duration of a session (minutes).
Exercise History questionnaire, part 2 (strength exercise) | Within 1 week following inclusion
  Strength: participation in strength training (yes/no).
  If yes: frequency (days/week) of strength training, further specified as:
  Per type of muscle-strengthening exercise (using weight machines/bodyweight exercises/resistance exercises/holistic exercises): frequency (days/week); duration (0/<10/10-20/21-30/31-40/41-50/51-60/>60 minutes); muscle groups trained (legs/hips/back/abdomen/chest/shoulders/arms). Intensity at which the abovementioned muscle-strengthening exercises will be performed (0-10, 0 being extremely light, 10 being extremely heavy).
  Other: room for further comments regarding exercise history
Other biomarker concentrations in blood | At day of inclusion
  creatinine concentration (µmol/L); estimated glomerular filtration rate (ml/min/1.73m2); total cholesterol concentration (mmol/L), HDL cholesterol concentration (mmol/L), LDL cholesterol concentration (mmol/L), albumin concentration (g/L), cardiac myosin binding protein C concentration(ng/ml).
  (HDL: high-density lipoprotein; LDL: low-density lipoprotein)

CONTACTS AND LOCATIONS:
Overall Officials: Thijs Eijsvogels, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data will be stored in the myDRE research environment platform (myDRE, anDREa BV (Digital Research Environment), Nijmegen, the Netherlands) for at least 20 years in a safe way adhering to the General Data Protection Regulation, Good Clinical Practice and Good Laboratory Practice guidelines. We will use standard software packages for data handling and statistical analyses (e.g. Castor EDC, SPSS, Microsoft Excel). In line with open science and the FAIR principles (Findable, Accessible, Interoperable and Reusable), data from the TREAT study will be made available for reuse upon reasonable request via the corresponding author.

REFERENCES:
- [Derived] Janssen SLJE, Lamers SK, Vroemen WHM, Denessen EJS, Berge K, Bekers O, Hopman MTE, Brink M, Habets J, Nijveldt R, Van Everdingen WM, Aengevaeren VL, Mingels AMA, Eijsvogels TMH. Cardiac troponin concentrations following exercise and the association with cardiovascular disease and outcomes: rationale and design of the prospective TREAT cohort study. BMJ Open Sport Exerc Med. 2024 Jun 13;10(2):e002070. doi: 10.1136/bmjsem-2024-002070. eCollection 2024. PMID 38882206

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT06295081/Prot_SAP_ICF_000.pdf